CLINICAL TRIAL: NCT07082504
Title: Effects of Physical Exercise Programs, Cognitive Stimulation, and Their Combination on Mobility, Cognitive Function, and Psychosocial Well-Being in Institutionalized Older Adults
Brief Title: Effects of Exercise, Cognitive Training, and Their Combination in Institutionalized Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Nuno Adriano Sousa Carvalho, Doctoral Program Student, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1379
Record Dates: First submitted 2025-06-27; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Aging; Institutionalized Older Adults; Cognitive Abilities; Mobility and Independence; Well-being/Quality of Life
Keywords: Physical Exercise; Cognitive Stimulation; Executive Function; Quality of Life; Elderly Adults; Physical Function; Dual-Task Training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical Exercise Group (Experimental): Participants will engage in moderate-intensity physical exercise sessions 3 times per week for 12 weeks (150 minutes per week), including balance, strength, and functional mobility exercises led by physiotherapists.
  Interventions: Behavioral: Physical Exercise Program
- Cognitive Stimulation Group (Experimental): Participants will attend 3 weekly sessions for 12 weeks, involving activities such as memory games, problem-solving tasks, orientation exercises, and attention training, led by a psychologist and a social educator.
  Interventions: Behavioral: Cognitive Stimulation Program
- Combined Intervention Group (Experimental): Participants will receive both the physical exercise and cognitive stimulation programs simultaneously, with the same weekly frequency and duration as the individual interventions.
  Interventions: Behavioral: Combined Physical Exercise and Cognitive Stimulation
- Control Group (No Intervention): Participants will continue their usual routines without structured physical or cognitive interventions. They will receive standard care provided by the institution.

INTERVENTIONS:
Behavioral: Physical Exercise Program — Participants will complete supervised moderate-intensity physical exercise sessions three times per week for 12 weeks (totaling 150 minutes per week). The program includes balance, flexibility, strength, and mobility exercises designed according to WHO and ACSM guidelines for older adults. Sessions are delivered in small groups by trained physiotherapists.
  Arms: Physical Exercise Group
Behavioral: Cognitive Stimulation Program — Participants will attend cognitive stimulation sessions three times per week for 12 weeks. Activities include memory games, attention tasks, puzzles, orientation exercises, and problem-solving strategies. The sessions are led by a psychologist and a trained social educator, in small groups.
  Arms: Cognitive Stimulation Group
Behavioral: Combined Physical Exercise and Cognitive Stimulation — Participants will receive both the physical exercise and cognitive stimulation interventions, conducted in parallel, over a 12-week period with three sessions per week. The combined program aims to improve physical and cognitive functions simultaneously and is delivered by a multidisciplinary team.
  Arms: Combined Intervention Group

SUMMARY:
The goal of this clinical trial is to learn if physical exercise, cognitive stimulation, or a combination of both can improve mobility, cognitive function, and psychosocial well-being in institutionalized older adults aged 65 and older. The main questions it aims to answer are:

* Does physical exercise improve strength, flexibility, balance, and mobility?
* Does cognitive stimulation improve executive function and mental state?
* Does combining both interventions provide greater benefits than either intervention alone?

Researchers will compare the physical exercise group, the cognitive stimulation group, and the combined group to a control group that receives no active intervention to see which approach leads to the most improvement.

Participants will:

* Take part in either physical exercise, cognitive stimulation, or both, 3 times per week for 12 weeks
* Complete assessments before the intervention, after 12 weeks, and again after 6 months
* Answer questionnaires and perform physical and cognitive tests to measure changes in health and well-being

ELIGIBILITY:
Inclusion Criteria:

* Individuals of both sexes.
* Age 65 years or older.
* Retired.
* Institutionalized for more than three months.
* Provide informed consent and agree to participate.

Exclusion Criteria:

* Lack of cooperation or cognitive capacity to participate.
* Diagnosis of dementia or Alzheimer's disease.
* Presence of acute medical conditions.
* Physical or cognitive impairments that prevent completion of study procedures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Functional Mobility Measured by the Timed Up and Go (TUG) Test at 12 Weeks | From baseline to the end of the intervention at 12 weeks.
  Functional mobility will be assessed using the Timed Up and Go (TUG) test. The participant is timed while rising from a chair, walking 3 meters, turning, returning, and sitting.
  Score: Time in seconds (lower values indicate better mobility).
Change from Baseline in Executive Function Assessed by the Stroop Test at 12 Weeks | From baseline to the end of the intervention at 12 weeks.
  Executive function will be assessed using the Stroop Color and Word Test, which evaluates attention, inhibition, and cognitive flexibility.
  Score: Time (seconds) and error count; lower values indicate better performance.
Change from Baseline in Quality of Life Measured by EQ-5D at 12 Weeks | From baseline to the end of the intervention at 12 weeks.
  The EQ-5D assesses five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  Score Range: -0.594 to 1. Higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Change in Balance Performance Measured by the Tinetti Performance Oriented Mobility Assessment (POMA) at 12 Weeks | From baseline to the end of the intervention at 12 weeks.
  Balance will be evaluated using the Tinetti POMA. Score Range: 0-28 points. Higher scores indicate better balance and lower risk of falls.
Change in Lower Body Strength Measured by the 30-Second Chair Stand Test at 12 Weeks | From baseline to the end of the intervention at 12 weeks.
  Participants will perform as many full stands as possible from a seated position in 30 seconds.
  Score: Number of stands. Higher numbers indicate better strength.
Change in Upper Body Strength Measured by the Arm Curl Test at 12 Weeks | From baseline to 12 weeks post-intervention.
  Upper body strength is assessed by the number of bicep curls in 30 seconds using a standardized weight (5 lbs for women, 8 lbs for men).
  Score: Number of repetitions. Higher scores indicate better strength.
Change in Grip Strength Measured by Hand Dynamometer at 12 Weeks | From baseline to 12 weeks post-intervention.
  Grip strength is measured using a handheld dynamometer. Score: Kilograms (kg). Higher scores indicate stronger grip.
Change in Sleep Quality Measured by the Pittsburgh Sleep Quality Index (PSQI) at 12 Weeks | From baseline to the end of the intervention at 12 weeks.
  SThe PSQI evaluates sleep duration, disturbances, latency, and overall quality. Score Range: 0-21. Lower scores indicate better sleep quality.
Change in Depressive Symptoms Measured by the Geriatric Depression Scale (GDS) at 12 Weeks | From baseline to the end of the intervention at 12 weeks.
  The GDS is a screening tool for depression in older adults. Score Range: 0-15. Lower scores indicate fewer depressive symptoms.
Change in Life Satisfaction Measured by the Satisfaction With Life Scale (SWLS) at 12 Weeks | From baseline to the end of the intervention at 12 weeks.
  The SWLS measures global cognitive judgments of satisfaction with life. Score Range: 5-35. Higher scores indicate greater life satisfaction.
Change in Functional Mobility Measured by the Timed Up and Go (TUG) Test at 6-Month Follow-Up | From the end of the intervention to 6 months follow-up.
  Follow-up assessment of mobility using the TUG test.
Change in Executive Function Measured by the Stroop Test at 6-Month Follow-Up | From baseline to the end of the intervention at 12 weeks.
  Follow-up assessment of executive function using the Stroop Test.
Change in Quality of Life Measured by the EQ-5D at 6-Month Follow-Up | From end of intervention to 6 months post-intervention.
  Follow-up assessment using the EuroQol-5 Dimension (EQ-5D).